CLINICAL TRIAL: NCT01073930
Title: A Randomized, Assessor-Blinded, Multi-Center Study Investigating the Efficacy, Safety and Tolerability of "Split-Dose" PicoPrep™ for Oral Administration Versus HalfLytely® for Colon Cleansing in Preparation for Colonoscopy
Brief Title: Investigation of PicoPrep Versus HalfLytely for Bowel Preparation for Colonoscopy - Split Dose PicoPrep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009-01
Record Dates: First submitted 2010-02-22; First posted 2010-02-23 (Estimated); Results first posted 2012-09-11 (Estimated); Last update posted 2013-02-12 (Estimated); Status verified 2013-02

CONDITIONS: Bowel Preparation
Keywords: Bowel Preparation; Colonoscopy
MeSH Terms: interventions — picosulfate sodium; Bisacodyl

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PICOPREP (Experimental): "Split Dose" method and consists of two separate doses: the first dose during the evening before the colonoscopy and the second dose the next day, during the morning prior to the colonoscopy.
  Interventions: Drug: PicoPrep
- HalfLytely (Active Comparator): HalfLytely and Bisacodyl Tablets Bowel Prep Kit was used according to the approved labeled dosage and administration instructions. The two bisacodyl tablets were taken the day prior to the procedure and the HalfLytely was taken following the first bowel movement or 6 hours after the bisacodyl tablets.
  Interventions: Drug: HalfLytely; Drug: bisacodyl

INTERVENTIONS:
Drug: PicoPrep — PICOPREP (sodium picosulfate, magnesium oxide and citric acid) powder for oral solution consisted of 2 pouches of powder administered in a divided dose. Each PICOPREP pouch was reconstituted by mixing the contents in a cup with 5 ounces of cold water. The first pouch was taken between 5:00 PM and 9:00 PM the evening prior to the colonoscopy procedure. Subjects were to consume five (5) 8-ounce glasses of clear liquids over the next few hours. The second pouch was taken approximately 5 hours before but no more than 9 hours prior to the colonoscopy procedure. Subjects were to consume three (3) 8-ounce glasses of clear liquids.
  Other Names: PicoPrep™; Prepopik™
  Arms: PICOPREP
Drug: HalfLytely — HalfLytely contains polyethylene glycol electrolyte solution (PEG-EL), sodium chloride, sodium bicarbonate and potassium chloride. The day prior to the colonoscopy procedure and after the first bowel movement or after 6 hours following administration of the bisacodyl tablets, whichever occurred first, subjects were to drink the 2 liter HalfLytely at a rate of one 8-ounce glass every 10 minutes. The entire solution was to be consumed.
  Arms: HalfLytely
Drug: bisacodyl — Two 5 mg bisacodyl tablets were taken in the afternoon on the day prior to the colonoscopy procedure.
  Arms: HalfLytely

SUMMARY:
Subjects undergoing an elective complete colonoscopy will randomly receive either PicoPrep: 2-sachets for oral solution in two divided doses given a night before (first dose - sachet) and approximately 5 hours prior to procedure (second dose - sachet) or HalfLytely: for oral solution and two 5 mg Bisacodyl tablets, given the day before the procedure to evaluate its effectiveness, tolerability and safety.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 to 80 years, inclusive, being scheduled to undergo elective colonoscopy
* Female patients should be post menopausal (women ≥ 45yrs with no menstrual period for at least 12 months without an alternative medical cause), be surgically sterile, or be using medically approved contraception, throughout the trial period
* Females of childbearing potential must undergo a pregnancy test at screening and again at randomization
* Subjects must have had more than or equal to 3 spontaneous bowel movements per week for one month prior to the colonoscopy
* Subjects should be willing, able and competent to complete the entire procedure and to comply with study instructions
* Written informed consent obtained prior to study

Exclusion Criteria:

* Acute surgical abdominal conditions (e.g. acute obstruction or perforation, etc.)
* Active (acute/exacerbation of/severe/uncontrolled) Inflammatory Bowel Disease (IBD)
* Any prior colorectal surgery, excluding appendectomy, hemorrhoid surgery or prior endoscopic procedures
* Colon disease (history of colonic cancer, toxic megacolon, toxic colitis, idiopathic pseudo-obstruction, hypomotility syndrome)
* Ascites
* Gastrointestinal disorder (active ulcer, outlet obstruction, retention, gastroparesis, ileus)
* Upper gastrointestinal surgery (gastric resection, gastric banding, gastric by-pass)
* Uncontrolled angina and/or Myocardial Infarction (MI) within last 3 months, Congestive Heart Failure (CHF), or uncontrolled hypertension
* Renal insufficiency (serum creatinine and potassium must be within normal limits)
* Participation in an investigational study within 30 days prior to receiving study medication (or within 60 days for investigational drugs with an elimination half-life greater than 15 days)
* Any clinically significant laboratory value at the screening, including pre-existing electrolyte abnormality, based on clinical history that the Investigator feels may affect the study evaluation
* Hypersensitivity to active ingredients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 608 (Actual)
Dates: Start 2010-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development Support, Study Director — Ferring Pharmaceuticals
Locations (9):
- United States (9):
  - Clinical Research Associates, Huntsville, Alabama
  - Arkansas Gastroenterology, Sherwood, Arkansas
  - Connecticut Gastroenterology Institute, Bristol, Connecticut
  - Indiana University Hospital, Indianapolis, Indiana
  - Louisiana Research Center LLC, Shreveport, Louisiana
  - Piedmont Medical Research Associates, Winston-Salem, North Carolina
  - Hillmont GI, P.C., Flourtown, Pennsylvania
  - ClinSearch, Chattanooga, Tennessee
  - Blue Ridge Medical Research, Lynchburg, Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PICOPREP | HalfLytely
Started | 307 | 301
Safety Population (Treated) | 305 | 298
Intent to Treat Population | 304 (One treated participant did not have an efficacy assessment performed.) | 297 (One treated participant did not have an efficacy assessment performed.)
Completed | 304 | 295
Not Completed | 3 | 6
Not completed — Withdrawal by Subject | 3 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Noncompliance with study drug | 0 | 1
Not completed — Inadequate prep; unable to do procedure | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PICOPREP | HalfLytely | Total
Number analyzed (Participants) | 305 | 298 | 603
Age Continuous [Mean (Standard Deviation); unit: years] | 54.8 (10.04) | 55.7 (10.00) | 55.2 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 181 | 174 | 355
  Male | 124 | 124 | 248
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 5 | 12
  Not Hispanic or Latino | 298 | 293 | 591
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 36 | 27 | 63
  White | 265 | 268 | 533
  Other | 3 | 0 | 3
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (5.68) | 29.6 (6.34) | 29.5 (6.01)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Classified as Successes (Excellent and Good Ratings) According to the Aronchick Scale As Assessed by a Blinded Gastroenterologist
Description: Overall colon cleansing was assessed by a blinded gastroenterologist during the colonoscopy using the Aronchick scale. The Aronchick scale is a 4-step rating scale: inadequate, fair, good, and excellent. Excellent is defined as >90% of mucosa seen, mostly liquid stool, minimal suctioning needed for adequate visualization. Good is defined as >90% of mucosa seen, mostly liquid stool, significant suctioning needed for adequate visualization.
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 304 | 297
percentage of participants | 84.2 | 74.4
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Non-Inferiority or Equivalence — Non-inferiority was demonstrated if the 1-sided 97.5% CI for the treatment difference (PICOPREP minus HalfLytely) was >-9% for the percentage of responders. Superiority was demonstrated if the 1-sided 97.5% CI for treatment difference was >0%; Mean Difference (Net) = 9.8, 97.5% CI 1-sided [lower limit 3.4]

2. Secondary Outcome: Percentage of Participants Classified as Successes (Excellent, Good and Fair Ratings) According to the Ottawa Scale As Assessed by a Blinded Gastroenterologist
Description: Overall colon cleansing was assessed by a blinded gastroenterologist during the colonoscopy using the Ottawa scale, a 5-step rating scale: inadequate, poor, fair, good, and excellent. Excellent is defined as mucosal detail clearly visible; if fluid is present, it is clear and there is almost no stool residue. Good - some turbid fluid or stool residue but mucosal detail still visible; washing and suctioning is not necessary. Fair - turbid fluid or stool residue obscuring mucosal detail. However, mucosal detail becomes visible with suctioning and washing is not necessary.
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 304 | 297
percentage of participants
  Ascending colon | 89.5 | 78.8
  Mid colon | 92.4 | 85.9
  Recto-sigmoid colon | 92.4 | 87.2
  Overall: ascending, mid, and recto-sigmoid colon | 86.8 | 75.4
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Ascending colon comparison; Test type: Non-Inferiority or Equivalence — If the lower bound of the 97.5% confidence interval exceeds -9.0% then PicoPrep will be declared non-inferior to HalfLytely. If the non-inferiority test is satisfied then a test for superiority will be performed by comparing the lower bound of the 97.5% confidence interval with 0.0%. If the lower bound of the confidence interval is above 0.0% then superiority will be declared; Mean Difference (Net) = 10.7, 97.5% CI 1-sided [lower limit 4.9]
Statistical Analysis 2: Comparison: PICOPREP vs HalfLytely; Mid colon comparison; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Net) = 6.6, 97.5% CI 1-sided [lower limit 1.6]
Statistical Analysis 3: Comparison: PICOPREP vs HalfLytely; Recto-sigmoid colon comparison; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Net) = 5.2, 97.5% CI 1-sided [lower limit 0.4]
Statistical Analysis 4: Comparison: PICOPREP vs HalfLytely; Overall: Ascending, mid, and recto-sigmoid colon comparison; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 2, analysis 1]; Mean Difference (Net) = 11.4, 97.5% CI 1-sided [lower limit 5.2]

3. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: How Easy or Difficult Was It To Consume the Study Drug?
Description: Participants answered the question above on Day 2 prior to the colonoscopy procedure. Answers were on a 5-point scale: very easy, easy, tolerable, difficult, very difficult
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed. Three participants either did not complete the questionnaire or did not answer this question.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 302 | 296
percentage of participants
  Very easy | 57.9 | 8.1
  Easy | 31.5 | 20.9
  Tolerable | 9.6 | 47.0
  Difficult | 1.0 | 14.9
  Very difficult | 0 | 9.1
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: Were You Able to Consume the Entire Prep As Instructed?
Description: Participants answered the question above on Day 2 prior to the colonoscopy procedure. Answers were on a 2-point scale: yes, no
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed. Two participants either did not complete the questionnaire or did not answer this question.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 303 | 296
percentage of participants
  Yes | 99.0 | 89.9
  No | 1.0 | 10.1
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Fisher Exact

5. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: Please Describe Your Overall Experience With the Study Preparation
Description: Participants answered the question above on Day 2 prior to the colonoscopy procedure. Answers were on a 5-point scale: Excellent, Good, Fair, Poor, Bad
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed. Four participants either did not complete the questionnaire or did not answer this question.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 301 | 296
percentage of participants
  Excellent | 46.8 | 16.6
  Good | 45.2 | 42.9
  Fair | 6.6 | 28.7
  Poor | 1.0 | 7.1
  Bad | 0.3 | 4.7
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: The Taste of This Study Preparation Was
Description: Participants answered the question above on Day 2 prior to the colonoscopy procedure. Answers were on a 5-point scale: Excellent, Good, Tolerable, Poor, Bad
Time Frame: Day 2
Population: Intent-to-treat population of randomized and treated participants with efficacy assessments performed. One participant either did not complete the questionnaire or did not answer this question.
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 303 | 297
percentage of participants
  Excellent | 23.4 | 2.7
  Good | 50.5 | 18.9
  Tolerable | 25.7 | 56.2
  Poor | 0.3 | 13.1
  Bad | 0 | 9.1
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: Would You Ask Your Doctor for This Preparation Again if You Need Another Colonoscopy in the Future?
Description: as for outcome 4
Time Frame: Day 2
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 302 | 296
percentage of participants
  Yes | 96.0 | 54.7
  No | 4.0 | 45.3
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Fisher Exact

8. Secondary Outcome: Percentage of Participants' Responses to the Acceptability and Tolerability Questionnaire: Would You Refuse the Same Preparation Again if it Were to be Prescribed to You in the Future?
Description: as for outcome 4
Time Frame: Day 2
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 301 | 296
percentage of participants
  Yes | 1.7 | 13.5
  No | 98.3 | 86.5
Statistical Analysis 1: Comparison: PICOPREP vs HalfLytely; Test type: Superiority or Other; p < 0.0001, Fisher Exact

9. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: Counts of participants who had TEAEs are summarized in a variety of categories. Severity and relatedness to study drug are in the opinion of the investigator. Severity is rated on a 3-point scale: mild (awareness of signs or symptoms, but no disruption of usual activity), moderate (event sufficient to affect usual activity), and severe (inability to work or perform usual activities). Only severe TEAEs are summarized. Relatedness is assessed on a 4-point scale: unrelated, unlikely, possibly and probably. Both possibly and probably answers are reported as 'related' to study medication.
Time Frame: up to one month
Population: Safety population of participants who were treated.
Measure: Number; unit: participants
Arm/Group | PICOPREP | HalfLytely
Number analyzed (Participants) | 305 | 298
participants
  Any TEAE | 211 | 217
  Death | 0 | 0
  Serious AE | 1 | 2
  TEAEs leading to discontinuation of study drug | 0 | 1
  Severe TEAEs | 2 | 6
  Related TEAEs | 19 | 26

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs occurring from Day 1 up to one month
Arm/Group | PICOPREP | HalfLytely
Serious Adverse Events (participants affected / at risk) | 1/305 | 2/298
Other Adverse Events (participants affected / at risk) | 166/305 | 177/298
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PICOPREP (N=305) | HalfLytely (N=298)
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PICOPREP (N=305) | HalfLytely (N=298)
Colonic polyp (Gastrointestinal disorders) | 52 | 51
Diverticulum (Gastrointestinal disorders) | 60 | 72
Diverticulum intestinal (Gastrointestinal disorders) | 11 | 16
Haemorrhoids (Gastrointestinal disorders) | 54 | 59
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 56 | 51

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review the draft manuscript prior to publication and can request delay of publication where any contents are deemed patentable by the sponsor or confidential to the sponsor. Comments will be given within four weeks from receipt of the draft manuscript. Additional time may be required to allow Ferring to seek patent protection of the invention.